CLINICAL TRIAL: NCT04358978
Title: A Novel Approach to Posterior Mesh Fixation in Laparoscopic Sacral Colpopexy: a Randomized Control Trial
Brief Title: A Novel Approach to Posterior Mesh Fixation in Laparoscopic Sacral Colpopexy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Catholic University of the Sacred Heart (Other)
Collaborators: Miulli General Hospital (Other)
Responsible Party: Principal Investigator, Maurizio Guido, principal investigator, Director of gynaecologic and obstetric department, Catholic University of the Sacred Heart
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Ospedale "F. Miulli"
Record Dates: First submitted 2020-04-21; First posted 2020-04-24 (Actual); Last update posted 2020-07-24 (Actual); Status verified 2020-07

CONDITIONS: Pelvic Organ Prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- posterior mesh no attachment (Active Comparator): laparoscopic sacral colpopexy with no fixation of posterior mesh
  Interventions: Procedure: laparoscopic sacral colpopexy with posterior mesh no attachment
- posterior mesh attachment (Active Comparator): laparoscopic sacral colpopexy with fixation of posterior mesh by suture
  Interventions: Procedure: laparoscopic sacral colpopexy with posterior mesh attachment

INTERVENTIONS:
Procedure: laparoscopic sacral colpopexy with posterior mesh no attachment — pelvic organ prolapse correction with laparoscopic sacralcolpopexy with no attachement of posterior mesh
  Arms: posterior mesh no attachment
Procedure: laparoscopic sacral colpopexy with posterior mesh attachment — pelvic organ prolapse correction with laparoscopic sacralcolpopexy with the attachement of posterior mesh to vagina
  Arms: posterior mesh attachment

SUMMARY:
This randomized controlled study is designed to test the non inferiority of no attachment of posterior mesh compared to fixation of posterior mesh to the vagina in laparoscopic sacral colpopexy in terms of anatomical correction of the prolapse, post-operative and long term morbidity and rate of recurrence.

ELIGIBILITY:
Inclusion Criteria:

-patients who required surgical treatment for symptomatic pelvic organ prolapse stage ≥ 2 with or without stress urinary incontinence

Exclusion Criteria:

* Age > 75 years
* Severe cardiovascular or respiratory disease
* Pregnancy

Max Age: 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-04-23 (Actual); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
correction of pelvic organ prolapse | 1 year
  number of women with correction of prolapse mesured in S POP-Q stage during FU visit

SECONDARY OUTCOMES:
rate of recurrence | 1 year
  number of women with de novo anterior or posterior or central prolapse
long term outcomes | 1 year
  number of women with nicturia, dysuria, obstructed defecation , urinary incontinence, pelvic pain

CONTACTS AND LOCATIONS:
Locations (1):
- ospedale regionale Miulli, Acquaviva delle Fonti, Bari, Italy